CLINICAL TRIAL: NCT05016453
Title: Long-term Efficacy of Percutaneous Tibial Nerve Stimulation for Faecal Incontinence and New Approach for Partial Responders
Brief Title: Long-term Efficacy of Percutaneous Tibial Nerve Stimulation Applied to Patients With Faecal Incontinence.
Acronym: PTNSLONG
Status: Completed | Type: Observational
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, Luis Sánchez Guillen, Clinical Professor Luis Sánchez-Guillén, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Other Study IDs: PTNSLONGTERMEFFICACY
Record Dates: First submitted 2021-07-06; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Faecal Incontinence
Keywords: percutaneous tibial nerve stimulation; anal physiology; faecal incontinence; partial response; long-term efficacy
MeSH Terms: conditions — Encopresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Percutaneous tibial nerve stimulation (PTNS) is an ambulatory therapy validated for patients with Faecal Incontinence (FI) refractory to conservative treatment with proved short and mid-term efficacy.

The investigators therefore aimed to evaluate the long-term efficacy of PTNS, considered 3 years of follow-up. The investigators also aimed to identify predictors of responses and suggest a new approach for partial responders.

DETAILED DESCRIPTION:
Prospective single-centre cohort of patients with FI treated with PTNS was analysed.

PTNS sessions were performed in three phases: weekly for three months in the first phase, biweekly for three months in the second phase, and monthly for six months in the third and final phase.

Clinical control at the end of each phase and an additional follow-up was performed at 36 months. Wexner score, faecal urgency, bowel habits and quality of life for FI were assessed.

Patients were categorized in three groups: optimal responders when there was an improvement in Wexner score > 50%; partial responders if the improvement in Wexner score was 25-50%; and non-responders, when the improvement of Wexner score was < 25%.

Optimal responders and partial responders progressed into successive phases, whereas non-responders abandoned PTNS and other treatment options were offered.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of faecal incontinence for more than 6 months, refractory to conservative treatment.

Exclusion Criteria:

* Anatomic injuries that require surgery.
* External anal sphincter lesion of > 180º.
* Unavailability to attend regularly outpatient clinic.
* Major psychologic or psychiatric comorbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years old, diagnosed with faecal incontinence (at least one or more episodes of faecal incontinence for more than 6 months) refractory to conservative treatment.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2010-01-08 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2021-04-24 (Actual)

PRIMARY OUTCOMES:
Change in faecal incontinence assessed by Wexner Score | Baseline compared to 3, 6, 12 and 36 months after start of PTNS
  Rate of patients with improvement in faecal incontinence assessed by Wexner score (Maximum punctuation: 20 being severe incontinence. Minimum punctuation: 0, no incontinence).

SECONDARY OUTCOMES:
Predictors of good long-term improvement in Wexner score | At 3, 6 and 12 months after start of PTNS
  Influence of previous obstetric or surgery history and duration of symptoms in the variation of Wexner score
Partial Responders | At 3, 6 and12 months after start of PTNS
  Incidence of patients with a decrease in Wexner score between 25 and 50% compared to initial value, and their performance in the long term

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Universitario de Elche, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Macmillan AK, Merrie AE, Marshall RJ, Parry BR. The prevalence of fecal incontinence in community-dwelling adults: a systematic review of the literature. Dis Colon Rectum. 2004 Aug;47(8):1341-9. doi: 10.1007/s10350-004-0593-0. PMID 15484348
- [Background] Maestre Y, Pares D, Vial M, Bohle B, Sala M, Grande L. [Prevalence of fecal incontinence and its relationship with bowel habit in patients attended in primary care]. Med Clin (Barc). 2010 Jun 12;135(2):59-62. doi: 10.1016/j.medcli.2010.01.031. Epub 2010 Apr 22. Spanish. PMID 20416902
- [Background] MacLennan AH, Taylor AW, Wilson DH, Wilson D. The prevalence of pelvic floor disorders and their relationship to gender, age, parity and mode of delivery. BJOG. 2000 Dec;107(12):1460-70. doi: 10.1111/j.1471-0528.2000.tb11669.x. PMID 11192101
- [Background] Johanson JF, Lafferty J. Epidemiology of fecal incontinence: the silent affliction. Am J Gastroenterol. 1996 Jan;91(1):33-6. PMID 8561140
- [Background] Madoff RD. Surgical treatment options for fecal incontinence. Gastroenterology. 2004 Jan;126(1 Suppl 1):S48-54. doi: 10.1053/j.gastro.2003.10.015. PMID 14978638
- [Background] Jarrett ME, Mowatt G, Glazener CM, Fraser C, Nicholls RJ, Grant AM, Kamm MA. Systematic review of sacral nerve stimulation for faecal incontinence and constipation. Br J Surg. 2004 Dec;91(12):1559-69. doi: 10.1002/bjs.4796. PMID 15455360
- [Background] Thin NN, Horrocks EJ, Hotouras A, Palit S, Thaha MA, Chan CL, Matzel KE, Knowles CH. Systematic review of the clinical effectiveness of neuromodulation in the treatment of faecal incontinence. Br J Surg. 2013 Oct;100(11):1430-47. doi: 10.1002/bjs.9226. PMID 24037562
- [Background] Gupta P, Ehlert MJ, Sirls LT, Peters KM. Percutaneous tibial nerve stimulation and sacral neuromodulation: an update. Curr Urol Rep. 2015 Feb;16(2):4. doi: 10.1007/s11934-014-0479-1. PMID 25630918
- [Background] Hidalgo-Pujol M, Andriola V, Jimenez-Gomez LM, Ostiz F, Espin E. Medium-term outcome of percutaneous tibial nerve stimulation in the treatment of fecal incontinence. Tech Coloproctol. 2018 Nov;22(11):875-879. doi: 10.1007/s10151-018-1892-0. Epub 2018 Dec 18. PMID 30565161
- [Background] Hotouras A, Ribas Y, Allison M, Murphy J. The CONFIDeNT trial. Lancet. 2016 Feb 13;387(10019):643-644. doi: 10.1016/S0140-6736(16)00281-6. No abstract available. PMID 26876707
- [Background] de la Portilla F, Laporte M, Maestre MV, Diaz-Pavon JM, Gollonet JL, Palacios C, Vazquez-Monchul JM, Garcia-Cabrera AM, Jimenez-Rodriguez RM, Sanchez Gil JM. Percutaneous neuromodulation of the posterior tibial nerve for the treatment of faecal incontinence - mid-term results: is retreatment required? Colorectal Dis. 2014 Apr;16(4):304-10. doi: 10.1111/codi.12539. PMID 24617790
- [Background] Hotouras A, Murphy J, Walsh U, Allison M, Curry A, Williams NS, Knowles C, Chan CL. Outcome of percutaneous tibial nerve stimulation (PTNS) for fecal incontinence: a prospective cohort study. Ann Surg. 2014 May;259(5):939-43. doi: 10.1097/SLA.0b013e3182a6266c. PMID 23979291
- [Background] Munoz-Duyos A, Lagares-Tena L, Vargas-Pierolas H, Rodon A, Navarro-Luna A. High-resolution circuit for the diagnosis of faecal incontinence. Patient satisfaction. Cir Esp. 2017 May;95(5):276-282. doi: 10.1016/j.ciresp.2017.04.012. Epub 2017 Jun 8. English, Spanish. PMID 28602392
- [Background] Rockwood TH, Church JM, Fleshman JW, Kane RL, Mavrantonis C, Thorson AG, Wexner SD, Bliss D, Lowry AC. Fecal Incontinence Quality of Life Scale: quality of life instrument for patients with fecal incontinence. Dis Colon Rectum. 2000 Jan;43(1):9-16; discussion 16-7. doi: 10.1007/BF02237236. PMID 10813117
- [Background] Hotouras A, Thaha MA, Allison ME, Currie A, Scott SM, Chan CL. Percutaneous tibial nerve stimulation (PTNS) in females with faecal incontinence: the impact of sphincter morphology and rectal sensation on the clinical outcome. Int J Colorectal Dis. 2012 Jul;27(7):927-30. doi: 10.1007/s00384-011-1405-3. Epub 2012 Jan 25. PMID 22274577
- [Background] Lemon SC, Roy J, Clark MA, Friedmann PD, Rakowski W. Classification and regression tree analysis in public health: methodological review and comparison with logistic regression. Ann Behav Med. 2003 Dec;26(3):172-81. doi: 10.1207/S15324796ABM2603_02. PMID 14644693
- [Background] Shafik A, Ahmed I, El-Sibai O, Mostafa RM. Percutaneous peripheral neuromodulation in the treatment of fecal incontinence. Eur Surg Res. 2003 Mar-Apr;35(2):103-7. doi: 10.1159/000069399. PMID 12679620
- [Background] Queralto M, Portier G, Cabarrot PH, Bonnaud G, Chotard JP, Nadrigny M, Lazorthes F. Preliminary results of peripheral transcutaneous neuromodulation in the treatment of idiopathic fecal incontinence. Int J Colorectal Dis. 2006 Oct;21(7):670-2. doi: 10.1007/s00384-005-0068-3. Epub 2005 Dec 6. PMID 16331464
- [Background] Govaert B, Pares D, Delgado-Aros S, La Torre F, Van Gemert WG, Baeten CG. A prospective multicentre study to investigate percutaneous tibial nerve stimulation for the treatment of faecal incontinence. Colorectal Dis. 2010 Dec;12(12):1236-41. doi: 10.1111/j.1463-1318.2009.02020.x. PMID 19674028
- [Background] Thomas GP, Dudding TC, Bradshaw E, Nicholls RJ, Vaizey CJ. A pilot study to compare daily with twice weekly transcutaneous posterior tibial nerve stimulation for faecal incontinence. Colorectal Dis. 2013 Dec;15(12):1504-9. doi: 10.1111/codi.12428. PMID 24118972
- [Background] Arroyo Fernandez R, Avendano Coy J, Ando Lafuente S, Martin Correa M feminineT, Ferri Morales A. Posterior tibial nerve stimulation in the treatment of fecal incontinence: a systematic review. Rev Esp Enferm Dig. 2018 Sep;110(9):577-588. doi: 10.17235/reed.2018.5007/2017. PMID 30168339
- [Background] Pena Ros E, Parra Banos PA, Benavides Buleje JA, Munoz Camarena JM, Escamilla Segade C, Candel Arenas MF, Gonzalez Valverde FM, Albarracin Marin-Blazquez A. Short-term outcome of percutaneous posterior tibial nerve stimulation (PTNS) for the treatment of faecal incontinence. Tech Coloproctol. 2016 Jan;20(1):19-24. doi: 10.1007/s10151-015-1380-8. PMID 26499791
- [Background] Lopez-Delgado A, Arroyo A, Ruiz-Tovar J, Alcaide MJ, Diez M, Moya P, Santos J, Calpena R. Effect on anal pressure of percutaneous posterior tibial nerve stimulation for faecal incontinence. Colorectal Dis. 2014 Jul;16(7):533-7. doi: 10.1111/codi.12628. PMID 24674305
- [Background] Leroi AM, Siproudhis L, Etienney I, Damon H, Zerbib F, Amarenco G, Vitton V, Faucheron JL, Thomas C, Mion F, Roumeguere P, Gourcerol G, Bouvier M, Lallouche K, Menard JF, Queralto M. Transcutaneous electrical tibial nerve stimulation in the treatment of fecal incontinence: a randomized trial (CONSORT 1a). Am J Gastroenterol. 2012 Dec;107(12):1888-96. doi: 10.1038/ajg.2012.330. Epub 2012 Oct 2. PMID 23032981